CLINICAL TRIAL: NCT00055289
Title: Role of Multimodal Areas for Sensory-To-Motor Processing
Brief Title: Brain Use of Sensory Information to Generate Movement
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030112; 03-N-0112
Record Dates: First submitted 2003-02-22; First posted 2003-02-24 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-01

CONDITIONS: Healthy
Keywords: Transcranial Magnetic Stimulation; Counting; Sensorimotor Integration; Superior Temporal Cortex; Dorsal Premotor Cortex; Healthy Volunteer; HV

SUMMARY:
This study will use transcranial magnetic stimulation (TMS) to investigate functions of brain regions that may use information from sensory organs, such as the eyes or ears, to generate movements.

For TMS, a wire coil is held over the scalp. A brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. This may cause a pulling sensation on the skin under the coil and twitching in muscles of the face, arm, or leg. During the stimulation, the participant may be asked to tense certain muscles slightly or perform other simple actions.

Healthy normal volunteers 18 years of age and older may be eligible for this study. Individuals with a history of neuropsychiatric disorders, brain lesions such as tumors, stroke, or trauma, or a history of significant medical disorders, such as cancer, may not participate. Candidates will be screened with a medical history, brief physical examination, and questionnaire.

Participants will be presented a sequence of shapes (circles, rectangles, and triangle) and will count the number of a specified shape. Each number is assigned to a corresponding response button. The subject will push the appropriate button with the corresponding finger. During these experiments, the scalp will be stimulated by TMS. Each set of TMS measurements will take up to 3-1/2 hours.

DETAILED DESCRIPTION:
The role of multimodal brain regions for sensory-to-motor processing is not well understood. In our recent neuroimaging study with fMRI, we found that multimodal areas such as the right superior temporal cortex and right dorsal premotor cortex were activated during sensory instructed movements. These regions might contribute to extract common features or concepts from sensory stimuli, but we do not have firm experimental evidence yet. In order to investigate the functional roles of multimodal brain regions further, we propose to apply a transcranial magnetic stimulation (TMS) technique. TMS can create transient brain lesions allowing functional mapping of cortical regions. In this protocol, by stimulating the multimodal areas using TMS, we will determine the functional role of these areas.

ELIGIBILITY:
INCLUSION CRITERIA:

Forty normal volunteers will be included. Normal volunteers would be recruited from people who are registered as HMCS Normal Volunteers. All subjects participating in this study should have a valid Clinical Center Medical Record Number. Procedures for the experiment will follow the Standard Operating Procedures of HMCS TMS group.

EXCLUSION CRITERIA:

Contraindications for TMS;

Magnetic stimulation will not be performed in people who have pacemakers, implanted pumps or stimulators, or have metal objects inside the eye or skull. If the participants find the procedures too uncomfortable, they may discontinue the study at any time. Brain functions at a development stage are out of scope of this particular experiment. In this study, subjects 18 years or older will be included.

Contraindications for MRI;

Pacemakers, brain stimulators, dental implants or metallic braces, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, insulin pump, or shrapnel fragments. Welders and metal workers are also at risk for injury because of possible small metal fragments in the eye which they may be unaware. Subjects will be screened for these contraindications prior to the study.

Subjects with previous or current neuropsychiatric disorders will be excluded. Patients with MRI findings consistent with organic brain lesions such as brain tumors, stroke, or trauma will be excluded. Subjects not capable of giving informed consent will be excluded.

We will not scan pregnant women with MRI because safety of high magnetic field to fetus is not established. Therefore, we will administer a urine pregnancy test for any female subject of childbearing potential prior to MRI scan. Brain functions at a developmental stage are out of scope of this particular experiment. In this study, subjects aged 18 years or older will be included.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2003-02; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bremmer F, Schlack A, Shah NJ, Zafiris O, Kubischik M, Hoffmann K, Zilles K, Fink GR. Polymodal motion processing in posterior parietal and premotor cortex: a human fMRI study strongly implies equivalencies between humans and monkeys. Neuron. 2001 Jan;29(1):287-96. doi: 10.1016/s0896-6273(01)00198-2. PMID 11182099
- [Background] Calvert GA. Crossmodal processing in the human brain: insights from functional neuroimaging studies. Cereb Cortex. 2001 Dec;11(12):1110-23. doi: 10.1093/cercor/11.12.1110. PMID 11709482
- [Background] Chen R, Classen J, Gerloff C, Celnik P, Wassermann EM, Hallett M, Cohen LG. Depression of motor cortex excitability by low-frequency transcranial magnetic stimulation. Neurology. 1997 May;48(5):1398-403. doi: 10.1212/wnl.48.5.1398. PMID 9153480